CLINICAL TRIAL: NCT00470769
Title: Color-Doppler Ultrasonography vs 99mTc-DTPA Scintigraphy to Assess the Renal Blood Flow
Brief Title: The Efficacy of Color-Doppler Ultrasonography to Assess the Renal Blood Flow With the Estimation of GFR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Other Study IDs: CR-UR-00001
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Hypertension; Renal Failure
Keywords: Color-Doppler Ultrasonography; Renal scintigraphy; Kidney failure; GFR
MeSH Terms: conditions — Hypertension; Renal Insufficiency

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Color-Doppler Ultrasound, 99mTc-DTPA scintigraphy

SUMMARY:
It is generally assumed that renal blood flow is symmetric in the absence of renal artery stenosis. The importance of studying the function of both kidneys separately is because it cannot be assumed that they are functionally equal.The aim of the present study is to evaluate whether this is really in patients with essential hypertension and/or moderate kidneys loss.

DETAILED DESCRIPTION:
To validate color Doppler ultrasonography of renal arteries for the assessment of renal blood flow (RBF), we comparing left and right RBF estimates and their sum (total RBF) by echo-Doppler with data obtained by 99mTc-DTPA scintigraphy in 50 patients with hypertension and/or moderate renal failure, compared with 30 normal control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension
* Patients with moderate renal insufficiency
* Normal subjects

Exclusion Criteria:

* Patients with solitary kidney function
* Patients with renal artery stenosis
* Patients underwent renal angioplasty and stenting

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2006 (Estimated)
Dates: Start 2006-09; Study Completion 2007-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Cianci, MD, Principal Investigator — Department Of Clinic Medicine, Chair of Nephrology; Giorgio Fuiano, MD, Study Director — University of Catanzaro
Locations (3):
- Italy (3):
  - Giorgio Fuiano, Catanzaro
  - University of Rome La Sapienza, Roma
  - Rosario Cianci, Rome